CLINICAL TRIAL: NCT01343459
Title: Hypofractionated Whole-Breast Irradiation Preceded by Intra-Operative Radiotherapy With Electrons as Anticipated Boost HIOB A New Option in Breast-Conserving Treatment for Operated Breast Cancer Stages I and II
Brief Title: Intra-Operative Electron Boost and Hypofractionated Whole-Breast Irradiation During Breast-conserving Treatment (BCT)
Acronym: HIOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Medical University (Other)
Collaborators: LKH Klagenfurt (Other); Poznan University of Medical Sciences (Other); San Filippo Neri General Hospital (Other); Avera McKennan Hospital & University Health Center (Other); St. Luke's Hospital ,Cedar Rapids, US (Unknown); A.O.U. San Giovanni Battista di Torino, Italy (Other); IRCCS Cancer Referral Center of Basilicata (Other); Heinrich-Heine University, Duesseldorf (Other); St. Elisabeth-Hospital Köln-Hohenlind, Germany (Unknown); S.C. Radiotherapia Aziendale Umbria, Italy (Other); Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other); Fondazione Salvatore Maugeri (Other); Marien Hospital Düsseldorf (Other); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); Philipps University Marburg (Other); Istituti Tumori Giovanni Paolo II (Network); University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gerd Fastner, Assoc. Prof., MD, Paracelsus Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIORT - 01; ISIORT 01 (Other: ISIORT)
Record Dates: First submitted 2011-04-26; First posted 2011-04-28 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Local Neoplasm Recurrence; Toxicity
Keywords: Hypofractionated Whole breast irradiation; Hypofractionated Whole breast irradiation long term results; Breast conserving therapy; IORT with electrons in breast cancer; IOERT as anticipated Boost; IOERT and hypofractionated whole breast irradiation
MeSH Terms: conditions — Neoplasm Recurrence, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IOERT followed by hypofractionated WBRT (Experimental): HIOB: IOERT of 11.1 Gy followed by WBRT with 15 times 2.7 Gy per fraction.
  Interventions: Radiation: HIOB

INTERVENTIONS:
Radiation: HIOB — IOERT single shot as a boost followed by hypofractionated WBRT (HIOB)
  * IOERT is performed on mobile or fixed linacs
  * Reference dose: 11 Gy specified as maximum dose, with a minimum target volume dose of 90% encompassing the PTV (i.e. 10 Gy).
  WBRT
  * must start within day 36- 56 postoperatively (week 6 - 8 p.o.) in case of adjuvant hormonal treatment (or no further tumor specific medication)
  * In case of adjuvant chemotherapy, a time - gap between IOERT and WBRT up to 9 months is allowed.
  * Single reference dose per fraction: 2,7 Gy (ICRU)
  * Number of fractions: 15, Number of fractions per week: 5
  * Total WBRT dose: 40,5 Gy

SUMMARY:
Title:

HIOB - Hypofractionated Whole-Breast Irradiation preceded by Intraoperative Radiotherapy with Electrons as anticipated Boost ISIORT- 01

HIOB is defined as hypofractionated WBRT (40,5 Gy in 2,7 Gy per fraction) preceded by an Intraoperative Boost to the tumor bed ( 90 % reference dose of 10 Gy, 11,1 Gy Dmax IOERT).

Primary endpoint is the proof of superiority of a new treatment regimen.

The HIOB study concept is supposed to test the hypothesis whether such a combined schedule is superior (or iso-effective) towards "standard" RT in terms of local control and cosmetic outcome.

In the vast majority of all publications, annual and 5 year in-breast recurrence rates following BCT showed a clear dependency on patient age within the following boundaries (primary references):

Age > 50: Bartelink (standard): 0,7% (annual) 3,5% (5y) START B (best): 0,4 %(annual) 2,0% (5y)

Age 41-50: Bartelink (standard) 1,2% (annual) 6,0% (5y) Whelan (best) 0,72%(annual) 3,6% (5y)

Age ≥ 35-40 Bartelink (standard) 2% (annual) 10% (5y) Whelan (best) 0,72% (annual) 3,6% (5y)

long these three different age groups, benchmarking will be performed against the best published results following 'Golden Standard'RT, usually defined as conventionally fractionated WBRT with 50 Gy (25 x2) plus external tumor bed boost with 10-16 Gy electrons (5-8x2Gy).

Superiority is defined as going below the lower limit of the estimated 5 year local recurrence rate within the respective age group Inferiority is defined as crossing the respective upper limit .

Secondary endpoint:

Disease free survival

Tertiary endpoint: toxicity assessment (acute and late) including long term cosmetic evaluation

Study design and statistics:

* Prospective multicenter single-armed
* Sequential probability ratio test (SPRT)
* Separate analysis within three different age groups

Estimated Accrual time: strongly dependent on recruitment per year within the respective age group . Due to the statistical estimation of Szenario A and B the study will close after max. Time-period of 10 years in case of A or 6,4 years in case of B..

Principal investigators and study coordinators:

UC of Radiotherapy and Radio-Oncology UC of Special Gynecology and Breast Cancer Center Landeskrankenhaus Salzburg, Paracelsus University Clinics

DETAILED DESCRIPTION:
Study population:

See Points 4.1 und 4.2 Inclusion/Exclusion criteria of the entire protocol

Operation:

* Lumpectomy / segmentectomy / tumorectomy with sufficient safety margins (see above). Lymph node assessment must follow a sentinel node concept.
* Perioperative antibiotic prophylaxis is mandatory
* After IORT, radio-opaque clips have to be fixed at the tumor bed.

Histology: R0-Resection is mandatory

Chemotherapy:

neoadjuvant:allowed adjuvant: allowed.

There are no limitations towards special chemotherapeutic schemes and schedules.

Radiotherapy:

IOERT

* IOERT is performed on mobile or fixed linacs
* Reference dose: 11 Gy specified as maximum dose, with a minimum target volume dose of 90% encompassing the PTV (i.e. 10 Gy).

WBRT

* must start within day 36- 56 postoperatively (week 6 - 8 p.o.) in case of adjuvant hormonal treatment (or no further tumor specific medication)
* In case of adjuvant chemotherapy, a time - gap between IOERT and WBRT up to 9 months is allowed.
* Single reference dose per fraction: 2,7 Gy (ICRU)
* Number of fractions: 15, Number of fractions per week: 5
* Total WBRT dose: 40,5 Gy

RT of regional lymphatics: exclusion criterion

Diagnostics of Local recurrence:

* yearly mammographies,
* optional breast sonography, MRI
* LR has to be histologically confirmed

Follow-up screening for detection of metastases (minimum requirements):

* Chest X-Ray, optional
* abdominal sonography, optional
* lab tests incl. tumor markers, optional

Assessment of acute toxicity of WBRT according to CTC-toxicity Scoring-systems:

Assessment of late toxicity according to LENT-SOMA scoring-systems

Assessment of cosmetic outcome according to 5-point- Scoring System (vanLimbergen) starting before WBRT, including photo documentation in standardized positions

ELIGIBILITY:
Inclusion Criteria:

* Histological proven invasive breast carcinoma
* Age: ≥ 35 years
* Tumor stage T1-2
* nodal status: N0-1
* Freedom of surgical margins: R0 (both invasive and in situ component), that means no ink on tumors (invasive or in situ) (ago-online.de) .
* Also multifocal disease within the same quadrant with a maximum distance of < 5 cm
* all grades G1-G3
* Hormonal receptor and Her-2 status: no limitations
* Informed and undersigned consent

Exclusion Criteria:

* In-situ Carcinoma without invasive component
* Age < 35
* Tumor stage T3,4
* Nodal status >N1
* if irradiation of regional lymphatics is required
* R1
* Re-excision after IOERT
* Immediately secondary mastectomy (not due to recurrence).
* Multicentricity according to international definition: > 5 cm distance to each other
* previous radiotherapy to the involved breast
* Karnofsky Index < 70%
* Mixed connective tissue diseases including rheumatoid Polyarthritis, Thrombangitis obliterans
* Chronic pre-existent lung disease (Lung fibrosis, Pneumokoniosis, late-type Allergies like Farmer lung; Asthma bronchiale, severe Emphysema, COPD III *)
* Cardiac Co-Morbidity: clinically positive coronary vessel disease, St.p. myocardial infarction, pacemakers and/or defibrillators)
* Distant metastases
* breast size (PTV) > 2500 ml
* missing written consent
* observed pregnancy

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1464 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
5 year local recurrence rate: Sequential Probability Ratio Test | 10 years
  Sequential Probability Ratio Test

SECONDARY OUTCOMES:
Acute toxicity: CTC-toxicity Scoring-system;Late toxicity: LENT-SOMA scoring-systems | 10 years
  CTC-toxicity Scoring-System;LENT-SOMA scoring-systems

OTHER OUTCOMES:
Cosmesis | 10 years
  van Limbergen Scoring System

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Fastner, Assoc.Prof., Principal Investigator — Dep. of Radiotherapy and Radio-Oncology, Paracelsus Medical University Salzburg
Locations (1):
- Paracelsus private university; University Clinic of Radio-Oncology, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartelink H, Horiot JC, Poortmans P, Struikmans H, Van den Bogaert W, Barillot I, Fourquet A, Borger J, Jager J, Hoogenraad W, Collette L, Pierart M; European Organization for Research and Treatment of Cancer Radiotherapy and Breast Cancer Groups. Recurrence rates after treatment of breast cancer with standard radiotherapy with or without additional radiation. N Engl J Med. 2001 Nov 8;345(19):1378-87. doi: 10.1056/NEJMoa010874. PMID 11794170
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bentzen SM, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial B of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet. 2008 Mar 29;371(9618):1098-107. doi: 10.1016/S0140-6736(08)60348-7. Epub 2008 Mar 19. PMID 18355913
- [Background] Whelan TJ, Kim DH, Sussman J. Clinical experience using hypofractionated radiation schedules in breast cancer. Semin Radiat Oncol. 2008 Oct;18(4):257-64. doi: 10.1016/j.semradonc.2008.04.008. PMID 18725113
- [Background] Whelan TJ, Pignol JP, Levine MN, Julian JA, MacKenzie R, Parpia S, Shelley W, Grimard L, Bowen J, Lukka H, Perera F, Fyles A, Schneider K, Gulavita S, Freeman C. Long-term results of hypofractionated radiation therapy for breast cancer. N Engl J Med. 2010 Feb 11;362(6):513-20. doi: 10.1056/NEJMoa0906260. PMID 20147717
- [Background] Ivaldi GB, Leonardi MC, Orecchia R, Zerini D, Morra A, Galimberti V, Gatti G, Luini A, Veronesi P, Ciocca M, Sangalli C, Fodor C, Veronesi U. Preliminary results of electron intraoperative therapy boost and hypofractionated external beam radiotherapy after breast-conserving surgery in premenopausal women. Int J Radiat Oncol Biol Phys. 2008 Oct 1;72(2):485-93. doi: 10.1016/j.ijrobp.2007.12.038. Epub 2008 Apr 11. PMID 18407434
- [Background] START Trialists' Group; Bentzen SM, Agrawal RK, Aird EG, Barrett JM, Barrett-Lee PJ, Bliss JM, Brown J, Dewar JA, Dobbs HJ, Haviland JS, Hoskin PJ, Hopwood P, Lawton PA, Magee BJ, Mills J, Morgan DA, Owen JR, Simmons S, Sumo G, Sydenham MA, Venables K, Yarnold JR. The UK Standardisation of Breast Radiotherapy (START) Trial A of radiotherapy hypofractionation for treatment of early breast cancer: a randomised trial. Lancet Oncol. 2008 Apr;9(4):331-41. doi: 10.1016/S1470-2045(08)70077-9. Epub 2008 Mar 19. PMID 18356109
- [Background] Owen JR, Ashton A, Bliss JM, Homewood J, Harper C, Hanson J, Haviland J, Bentzen SM, Yarnold JR. Effect of radiotherapy fraction size on tumour control in patients with early-stage breast cancer after local tumour excision: long-term results of a randomised trial. Lancet Oncol. 2006 Jun;7(6):467-71. doi: 10.1016/S1470-2045(06)70699-4. PMID 16750496
- [Background] Yarnold J, Ashton A, Bliss J, Homewood J, Harper C, Hanson J, Haviland J, Bentzen S, Owen R. Fractionation sensitivity and dose response of late adverse effects in the breast after radiotherapy for early breast cancer: long-term results of a randomised trial. Radiother Oncol. 2005 Apr;75(1):9-17. doi: 10.1016/j.radonc.2005.01.005. Epub 2005 Mar 16. PMID 15878095
- [Background] Reitsamer R, Sedlmayer F, Kopp M, Kametriser G, Menzel C, Deutschmann H, Nairz O, Hitzl W, Peintinger F. The Salzburg concept of intraoperative radiotherapy for breast cancer: results and considerations. Int J Cancer. 2006 Jun 1;118(11):2882-7. doi: 10.1002/ijc.21727. PMID 16381011
- [Background] Reitsamer R, Peintinger F, Sedlmayer F, Kopp M, Menzel C, Cimpoca W, Glueck S, Rahim H, Kopp P, Deutschmann H, Merz F, Brandis M, Kogelnik H. Intraoperative radiotherapy given as a boost after breast-conserving surgery in breast cancer patients. Eur J Cancer. 2002 Aug;38(12):1607-10. doi: 10.1016/s0959-8049(02)00116-8. PMID 12142049
- [Background] Sedlmayer F, Fastner G, Merz F, Deutschmann H, Reitsamer R, Menzel C, Ciabattoni A, Petrucci A, Hager E, Willich N, Orecchia R, Valentini V; International Society of Intraoperative Radiotherapy. IORT with electrons as boost strategy during breast conserving therapy in limited stage breast cancer: results of an ISIORT pooled analysis. Strahlenther Onkol. 2007 Dec;183 Spec No 2:32-4. doi: 10.1007/s00066-007-2013-6. No abstract available. PMID 18167006
- [Background] Whelan T, MacKenzie R, Julian J, Levine M, Shelley W, Grimard L, Lada B, Lukka H, Perera F, Fyles A, Laukkanen E, Gulavita S, Benk V, Szechtman B. Randomized trial of breast irradiation schedules after lumpectomy for women with lymph node-negative breast cancer. J Natl Cancer Inst. 2002 Aug 7;94(15):1143-50. doi: 10.1093/jnci/94.15.1143. PMID 12165639